CLINICAL TRIAL: NCT00002532
Title: TREATMENT OF ADULT PATIENTS WITH RELAPSING ACUTE LYMPHOCYTIC LEUKEMIA, A MULTICENTER TRIAL
Brief Title: Combination Chemotherapy in Treating Patients With Relapsed or Refractory Acute Lymphocytic Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hannover Medical School (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: GER-ALL-REZ-02/92; CDR0000078432 (Registry Identifier: PDQ (Physician Data Query)); EU-93001
Record Dates: First submitted 1999-11-01; First posted 2004-02-16 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2002-03

CONDITIONS: Leukemia
Keywords: recurrent adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Filgrastim; Asparaginase; Cytarabine; Daunorubicin; Dexamethasone; Etoposide; Idarubicin; Ifosfamide; Leucovorin; Methotrexate; Prednisolone; Vindesine

INTERVENTIONS:
Biological: filgrastim
Drug: asparaginase
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: etoposide
Drug: idarubicin
Drug: ifosfamide
Drug: leucovorin calcium
Drug: methotrexate
Drug: prednisolone
Drug: vindesine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have relapsed or refractory acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxic effects and feasibility of high-dose cytarabine and idarubicin in patients with refractory or relapsed acute lymphocytic leukemia (ALL) after a complete remission (CR) of less than 18 months. II. Determine the response of patients with ALL in first relapse after a CR of 18 months or more treated with a 2-phase re-induction regimen comprising prednisolone, vindesine, daunorubicin, asparaginase, intrathecal (IT) cytarabine, IT dexamethasone, and IT methotrexate followed by prednisolone, ifosfamide, high-dose methotrexate, leucovorin calcium, etoposide, and cytarabine (with a dose-escalation study of etoposide and cytarabine). III. Compare the effectiveness of these 2 regimens administered to these patients with the regimen administered to historic controls (protocol GER-ALL-REZ- 01/88).

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified by center, duration of complete remission (CR) (less than 18 months vs 18 months or more), and refractory disease (yes vs no). Patients with refractory or relapsed disease after a CR of less than 18 months are treated on Regimen A. Patients in first relapse after a CR of 18 months or more are treated on Regimen B. Regimen A: Patients receive idarubicin IV over 30 minutes followed by cytarabine IV over 3 hours on days 1-3 and filgrastim (G-CSF) subcutaneously (SC) daily beginning on day 5 and continuing until blood counts recover. Regimen B (2-phase reinduction): Patients receive oral prednisolone on days 1-21; vindesine IV and daunorubicin IV on days 1, 8, and 15; asparaginase IV on days 7, 8, 14, and 15; and methotrexate intrathecally (IT), cytarabine IT, and dexamethasone IT on days 1 and 8. When blood counts recover, patients receive oral prednisolone and ifosfamide IV over 1 hour on days 1-4; high-dose methotrexate IV continuously on day 1 followed by standard leucovorin calcium rescue; etoposide IV over 1 hour followed at least 8 hours later by cytarabine IV over 3 hours on days 3 and 4; and G-CSF SC beginning on day 6 and continuing until blood counts recover. Cohorts of 6 patients or more receive escalating doses of etoposide and cytarabine until the maximum tolerated dose is determined.

PROJECTED ACCRUAL: Approximately 60 patients (30 per regimen) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of refractory or relapsed acute lymphocytic leukemia No isolated extramedullary relapse (e.g., testicular, CNS) Combined extramedullary and bone marrow relapse allowed No uncontrolled, severe leukemic complications, e.g.: Pneumonia with hypoxia Shock Cardiac failure Hemorrhage No refractoriness to platelet transfusion No unaspirable pleural effusions or ascites in patients with first relapse

PATIENT CHARACTERISTICS: Age: 15 to 65 Performance status: Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: See Disease Characteristics No uncontrolled bleeding Hepatic: No severe liver disease Renal: Creatinine clearance at least 60 mL/min in patients with first relapse after a complete remission of 18 months or more Cardiovascular: See Disease Characteristics No severe cardiac disease (e.g., congestive heart failure, myocardial infarction within the past 6 months, or severe arrhythmia) Pulmonary: See Disease Characteristics No severe pulmonary disease that would preclude aggressive chemotherapy Other: No hypersensitivity to E. coli proteins No severe neurologic or other disease that would preclude aggressive chemotherapy No severe psychiatric disease or other condition that would preclude study

PRIOR CONCURRENT THERAPY: Not specified

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-01

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Freund, MD, Study Chair — Klinik und Poliklinik fuer Innere Medizin - Universitaet Rostock
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Germany